CLINICAL TRIAL: NCT06958133
Title: The Effects of Postoperative Kinesio Taping on Pain, Range of Motion, and Edema in Weber Type B Lateral Malleolar Fractures: A Randomized Controlled Trial
Brief Title: Effects of Postoperative Kinesio Taping in Weber Type B Lateral Malleolar Fractures
Acronym: KT-WeberB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-WeberB-2025
Record Dates: First submitted 2025-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Ankle Fractures; Syndesmotic Injuries; Postoperative Rehabilitation
Keywords: ankle fractures, kinesiology
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Other): Standard postoperative rehabilitation without Kinesio taping.
  Interventions: Other: Standard Postoperative Rehabilitation
- Kinesio Taping Group (Other): Standard postoperative rehabilitation plus Kinesio taping application.
  Interventions: Other: Standard Postoperative Rehabilitation; Other: Kinesio Taping

INTERVENTIONS:
Other: Standard Postoperative Rehabilitation — Standard rehabilitation protocol after surgical fixation of Weber type B ankle fractures without Kinesio taping.
Other: Kinesio Taping — Kinesio taping applied over the surgical ankle to assist in reducing postoperative pain, swelling, and improving range of motion.
  Arms: Kinesio Taping Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of postoperative Kinesio taping on pain, range of motion, and edema in patients undergoing surgical fixation for Weber type B lateral malleolar fractures.

DETAILED DESCRIPTION:
Patients with Weber type B lateral malleolar fractures treated surgically were randomized into two groups: a control group receiving standard rehabilitation and an intervention group receiving additional Kinesio taping. Outcomes assessed included visual analog scale (VAS) pain scores, dorsiflexion range of motion, and circumferential edema measurements at 1, 7, and 28 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Patients diagnosed with isolated Weber type B lateral malleolar fractures requiring surgical fixation
* Surgery performed within 7 days of injury
* Written informed consent provided

Exclusion Criteria:

* Open fractures
* Associated fractures of the medial or posterior malleolus requiring fixation
* Polytrauma patients
* History of previous ankle fractures or surgeries on the affected side
* Neurological or vascular compromise of the affected limb
* Known allergy to adhesive materials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in pain levels assessed by Visual Analog Scale (VAS) at 4 weeks postoperatively | 28 days
  VAS scores ranging from 0 (no pain) to 10 (worst pain) measured at postoperative day 1, day 7, and day 28.

SECONDARY OUTCOMES:
Change in ankle dorsiflexion range of motion at 4 weeks, measured in degrees using a goniometer. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No